CLINICAL TRIAL: NCT05353075
Title: Effects of Sub-Occipital Muscle Inhibition Technique With and Without Hold Relax Agonist Contraction of Hamstrings on Pain, Disability and Craniovertebral Angle in Neck Pain Patients With Hamstring Tightness
Brief Title: Sub-Occipital MIT With and Without HR Agonist Contraction of Hamstrings in Neck Pain Patients With Hamstring Tightness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0133 Sumaiya
Record Dates: First submitted 2022-04-21; First posted 2022-04-29 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Neck Pain Patients With Hamstring Tightness
Keywords: Hamstring Muscles; Neck Pain; Muscle Tightness; PNF Stretching; Range of Motion
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub Occipital Muscle Inhibition (Other): Subjects in this group will receive only Sub Occipital Muscle Inhibition Technique and heating pad for 10 minutes.
  Interventions: Other: Sub Occipital Muscle Inhibition
- Sub Occipital Inhibition with Hold Relax Agonist Contraction (Experimental): Subjects in this group will receive Sub Occipital Inhibition and Hold Relax Agonist Contraction of hamstrings.
  Interventions: Other: Sub Occipital Muscle Inhibition; Other: Sub Occipital Inhibition with Hold Relax Agonist Contraction

INTERVENTIONS:
Other: Sub Occipital Muscle Inhibition — The therapist sits at the head end of the table, palms beneath the subject's head, pads of his fingertips on the posterior arch of the atlas, which will be palpated by the therapist between the external occipital protuberance and the spinous process of the axis vertebra. The therapist locates the gap between the occipital condyles and the spinous phase of the C2 vertebra with the middle and ring fingers of both hands the therapist then rests the base of the skull on his or her hands, with toward the therapist. The pressure will be held at the same level for four minutes until tissue relaxation will be achieved. The subject will be asked to keep his eyes closed during the SMI technique to prevent eye movements disturbing the Sub occipital muscle tone.
Other: Sub Occipital Inhibition with Hold Relax Agonist Contraction — Therapist will passively flex the lower extremity with knee extended to the end range of Hip Flexion. Once the end range of motion will attain the patient will apply a 10second isometric force against the therapist manual resistance. After the isometric contraction of hamstring the patient will ask to perform a concentric contraction of opposing muscle (hip flexors) for 10 seconds. As the patient performs the concentric contraction the therapist takes up the slack into any ROM that was gained keeping limb into new stretch position for 10-15 seconds and then rest for 5 seconds. Three repetitions of this technique will be performed on each subject.
  Arms: Sub Occipital Inhibition with Hold Relax Agonist Contraction

SUMMARY:
Hamstrings and Sub occipital muscles are part of the superficial back line of the myofascial chain which connects the neck to the lower extremity and the soft tissue in the cervical spine links the dura and sub occipital muscle fascia. Increased tension in one or other part of this myofascial chain disturbs the whole superficial back line and compromises the flexibility. The objective of this study is to determine the Effects of Sub-Occipital Muscle Inhibition technique (MIT) with and without Hold Relax (HR) Agonist Contraction of Hamstrings on Pain, Disability and Craniovertebral angle in Neck pain patients with Hamstring Tightness. This study will be a randomized controlled trial and will be conducted in Physiotherapy center of AL-Mahmood Welfare Foundation Sahiwal. This study will be completed in time duration of 10 months after the approval of synopsis and consecutive sampling technique will be used. A sample size of 34 will be randomly assigned into two groups. Group A will be given Sub Occipital Muscle Inhibition treatment while Group B will be given Sub occipital Muscle Inhibition and Hold Relax Agonist Contraction of hamstring. Each group will be given three sessions per week. Data will be collected from all participants before first session of treatment and after 6th session of treatment by using Numeric Pain Rating Scale (NPRS), Neck Disability Index (NDI), Cervical Range of motion (CROM), Craniovertebral Angle (CVA) and Active knee extension (AKE) test measurement.

ELIGIBILITY:
Inclusion Criteria:

Age 25-40 years Both Genders ( Male and Female) Neck Pain on NPRS ≥5 NDI score ≥14 ( Moderate disability) Active knee extension lag ≥30 and considered as tight hamstrings

Exclusion Criteria:

Acute Low back or Neck pain History of lumbar and cervical herniated disc and spinal stenosis History of cervical spine surgery and Trauma History of vascular disease in head and neck Progressive neurological deficit or Inflammatory condition ( such as peripheral neuropath, rheumatoid arthritis) History of abdominal or pelvic surgery in last 6 months

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 2 weeks
  The NPRS is an 11-point numerical scale used to measure average pain experience over 7 days, and ranges from 0 (no pain) to 11 (worst imaginable pain). NPRS is considered a valid and reliable scale for measures of pain intensity.
Bubble Inclinometer for Active Knee Extension test | 2 weeks
  For popliteal angle and cervical range of motion bubble inclinometer will be used in this study.
  In the Active knee extension test, the subjects knee will be extended with the subject will lying in the supine position and the hip joint flexed to 90°. This test has good validity and reliability (0.75)
Neck disability index | 2 weeks
  Urdu version of neck disability index will be used in this study.It consists of ten items related to pain intensity, headache, concentration and different physical activities (lifting, personal care, recreation, work, driving, reading and sleeping) with six possible responses per item. The score of each item ranges from 0 to 5. The highest total possible score is 50, and this score is converted to a percentage. Higher scores represent higher levels of disability. The NDI has been shown to be a valid and reliable questionnaire for patients with neck pain.
Image J software for Craniovertebral Angle | 2 weeks
  Craniovertebral angle will be measured by using a camera and Image J analysis software. For this purpose, patient will sit on a stool or chair in comfortable position, hands should be relaxed on thighs and feet on floor. A camera will set at I meter distance from patient and perpendicular to the height of patient's shoulder. The measuring evaluator attached two body markers, one on the tragus of ear and the other on the seventh spinous process. Patients will be asked to fix their gaze on a mark on the wall directly in front of them. Once the photograph was obtained, the CVA was used to measure the angle between a line extending from the tragus of the ear to C7 and the horizontal line passing through the C7 spinous process.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Al-Mahmood Welfare Foundation, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genebra CVDS, Maciel NM, Bento TPF, Simeao SFAP, Vitta A. Prevalence and factors associated with neck pain: a population-based study. Braz J Phys Ther. 2017 Jul-Aug;21(4):274-280. doi: 10.1016/j.bjpt.2017.05.005. Epub 2017 May 20. PMID 28602744
- [Background] Onat SS, Polat CS, Bicer S, Sahin Z, Tasoglu O. Effect of Dry Needling Injection and Kinesiotaping on Pain and Quality of Life in Patients with Mechanical Neck Pain. Pain Physician. 2019 Nov;22(6):583-589. PMID 31775405
- [Background] Kim BB, Lee JH, Jeong HJ, Cynn HS. Effects of suboccipital release with craniocervical flexion exercise on craniocervical alignment and extrinsic cervical muscle activity in subjects with forward head posture. J Electromyogr Kinesiol. 2016 Oct;30:31-7. doi: 10.1016/j.jelekin.2016.05.007. Epub 2016 May 24. PMID 27261928
- [Background] Cho SH, Kim SH, Park DJ. The comparison of the immediate effects of application of the suboccipital muscle inhibition and self-myofascial release techniques in the suboccipital region on short hamstring. J Phys Ther Sci. 2015 Jan;27(1):195-7. doi: 10.1589/jpts.27.195. Epub 2015 Jan 9. PMID 25642072
- [Background] Jeong ED, Kim CY, Kim SM, Lee SJ, Kim HD. Short-term effects of the suboccipital muscle inhibition technique and cranio-cervical flexion exercise on hamstring flexibility, cranio-vertebral angle, and range of motion of the cervical spine in subjects with neck pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2018;31(6):1025-1034. doi: 10.3233/BMR-171016. PMID 30248030
- [Background] Dhiman NR, Das B, Mohanty C, Singh OP, Gyanpuri V, Raj D. Myofascial release versus other soft tissue release techniques along superficial back line structures for improving flexibility in asymptomatic adults: A systematic review with meta-analysis. J Bodyw Mov Ther. 2021 Oct;28:450-457. doi: 10.1016/j.jbmt.2021.06.026. Epub 2021 Jun 16. PMID 34776177
- [Background] Kwon SH, Chung EJ, Lee J, Kim SW, Lee BH. The Effect of Hamstring Relaxation Program on Headache, Pressure Pain Threshold, and Range of Motion in Patients with Tension Headache: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Sep 27;18(19):10137. doi: 10.3390/ijerph181910137. PMID 34639438
- [Background] Jeong ED, Kim CY, Kim NH, Kim HD. Immediate effects of static and proprioceptive neuromuscular facilitation stretching of hamstring muscles on straight leg raise, craniovertebral angle, and cervical spine range of motion in neck pain patients with hamstring tightness: A prospective randomized controlled trial. J Back Musculoskelet Rehabil. 2022;35(2):429-438. doi: 10.3233/BMR-201840. PMID 34151831
- [Background] Joshi DG, Balthillaya G, Prabhu A. Effect of remote myofascial release on hamstring flexibility in asymptomatic individuals - A randomized clinical trial. J Bodyw Mov Ther. 2018 Jul;22(3):832-837. doi: 10.1016/j.jbmt.2018.01.008. Epub 2018 Feb 17. PMID 30100320
- [Background] Wilke J, Vogt L, Niederer D, Banzer W. Is remote stretching based on myofascial chains as effective as local exercise? A randomised-controlled trial. J Sports Sci. 2017 Oct;35(20):2021-2027. doi: 10.1080/02640414.2016.1251606. Epub 2016 Nov 7. PMID 27819537